CLINICAL TRIAL: NCT02374710
Title: Tibial Tunnel Placement for ACL Reconstruction: A Prospective, Randomized Clinical Trial
Brief Title: Tibial Tunnel Placement for ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17922
Record Dates: First submitted 2015-02-18; First posted 2015-03-02 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Complete Tear, Knee, Anterior Cruciate Ligament; Rupture of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL Reconstruction: Anterior Tunnel (Experimental): During surgery prior to ACL reconstruction, a line will be measured to indicate 35% of the anterior-to-posterior (front to back) distance of the proximal tibia. The tibial tunnel will be placed anterior (in front) of the 35% line.
  Interventions: Procedure: ACL Reconstruction: Anterior Tunnel
- ACL Reconstruction: Posterior Tunnel (Active Comparator): During surgery prior to ACL reconstruction, a line will be measured to indicate 35% of the anterior-to-posterior (front to back) distance of the proximal tibia. The tibial tunnel will be placed posterior (in back) of the 35% line.
  Interventions: Procedure: ACL Reconstruction: Posterior Tunnel

INTERVENTIONS:
Procedure: ACL Reconstruction: Anterior Tunnel — ACL reconstruction with anterior tibial tunnel placement in reference to a point measuring 35% of the anterior-posterior distance of the proximal tibia.
  Arms: ACL Reconstruction: Anterior Tunnel
Procedure: ACL Reconstruction: Posterior Tunnel — ACL reconstruction with posterior tibial tunnel placement in reference to a point measuring 35% of the anterior-posterior distance of the proximal tibia.
  Arms: ACL Reconstruction: Posterior Tunnel

SUMMARY:
Although extensive research has been carried out on Anterior Cruciate Ligament (ACL) femoral tunnel placement, very little attention has been given to the tibial tunnel. Researchers have suggested that the tibial tunnel be placed in the center of the ACL footprint, which they described as being approximately 43% of the way (anterior-to-posterior) across the proximal tibia at its widest extent. However, others have suggested that a more anterior placement may yield improved biomechanical and clinical results. The center of the ACL footprint and the posterior aspect of the anterior horn of the lateral meniscus does not yield tibial tunnel placement a consistent percentage of the way across the tibial plateau; therefore, guidelines should be based on intraoperative fluoroscopic measurements. However, the question remaining is what percentage of the anterior-to-posterior distance across the tibia is the ideal location for the tibial tunnel in ACL reconstruction. This study will help answer that question.

Patients with a diagnosed rupture of the ACL who are scheduled for surgical reconstruction will be considered for enrollment. Eligible patients will be allocated to one of two groups based on the location of the tibial tunnel (anterior vs. posterior) during the surgical procedure. In addition to a baseline (pre-operative) evaluation, participants will return for follow-up visits at 6, 12, and 24 months post-surgery. Follow up will be completed at 24 months.

The primary objective of this study is to collect subjective and objective measures of knee-related function in patients with an anterior vs. posterior placed tibial tunnel through 24 months postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Age at time of randomization: 16 - 50 years (skeletally mature)
* Primary, uncomplicated ACL reconstruction
* Autograft (STG or BPTB)

Exclusion Criteria:

* Multiple ligament knee injury (full thickness)
* Revision ACL reconstruction
* ACL reconstruction with allograft
* Meniscectomy > 75%
* Treatable articular cartilage lesions
* Diagnosis of tibiofemoral or patellofemoral osteoarthritis (Kellgren Lawrence grade > II)
* Valgus alignment on long-leg cassette (weight bearing line outside of joint center)
* Prior surgery in the ankles, knees, or hips
* Clinical evidence of hip disease
* Patellofemoral joint instability
* Significant patellar or tibiofemoral mal-alignment
* BMI > 35
* Type 1 Diabetes Mellitus
* Known connective tissue disorder (e.g. Ehlers-Danlos)
* Peripheral neuropathy
* Neurovascular/ circulatory disorder
* Any form of inflammatory arthritis (e.g. rheumatoid arthritis, gout, pseudogout, lupus, etc.)
* Significant co-morbid conditions as determined by the investigator (e.g. malignancy, renal, hepatic disease, etc.)
* Known or suspected psychological disorder

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Joint Evaluation | 24 months
  Subjective knee-specific function

SECONDARY OUTCOMES:
Knee Injury Outcome and Osteoarthritis Score (KOOS) | 24 months
  Subjective knee-specific function
Marx Activity Rating Scale | 24 months
  Subjective rating of physical activity
Visual Analog Scale (VAS) | 24 months
  Subjective pain
Quadriceps Strength | 24 months
  Thigh muscle strength assessment
Gait Analysis | 24 months
  Assessment of 3-dimensional movement patterns while walking
Knee Arthrometer (KT-1000) | 24 months
  Anterior knee laxity

OTHER OUTCOMES:
Knee Joint Range of Motion | 24 months
  Knee movement measured by goniometer
Thigh Circumference | 24 months
  Measure of your thigh using a tape measure
X-Ray (AP, lateral views) | 24 months
  X-ray of you knee

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Miller, M.D., Principal Investigator — University of Virginia; Joseph M Hart, Ph.D., Study Director — University of Virginia
Locations (1):
- University of Virginia, Department of Orthopedic Surgery, Division of Sports Medicine, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Staubli HU, Rauschning W. Tibial attachment area of the anterior cruciate ligament in the extended knee position. Anatomy and cryosections in vitro complemented by magnetic resonance arthrography in vivo. Knee Surg Sports Traumatol Arthrosc. 1994;2(3):138-46. doi: 10.1007/BF01467915. PMID 7584195
- [Result] Bedi A, Maak T, Musahl V, Citak M, O'Loughlin PF, Choi D, Pearle AD. Effect of tibial tunnel position on stability of the knee after anterior cruciate ligament reconstruction: is the tibial tunnel position most important? Am J Sports Med. 2011 Feb;39(2):366-73. doi: 10.1177/0363546510388157. Epub 2010 Dec 20. PMID 21173195
- [Result] Hatayama K, Terauchi M, Saito K, Higuchi H, Yanagisawa S, Takagishi K. The importance of tibial tunnel placement in anatomic double-bundle anterior cruciate ligament reconstruction. Arthroscopy. 2013 Jun;29(6):1072-8. doi: 10.1016/j.arthro.2013.02.003. Epub 2013 Apr 6. PMID 23571132

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT02374710/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02374710/ICF_001.pdf